CLINICAL TRIAL: NCT04902742
Title: Comparison of Treatment Outcomes in Chronic Coccygodynia Patients Treated With Ganglion Impar Blockade Versus Caudal Epidural Steroid Injection: A Prospective Randomized Comparison Study
Brief Title: Comparing the Treatment Outcomes of Two Interventional Pain Procedures in Chronic Coccygodynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09.2019.395
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Tailbone Disorders

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ganglion impar block group (Active Comparator): Fluoroscopy-guided ganglion impar block is applied to patients in this group.
  Interventions: Procedure: Fluoroscopy-guided ganglion impar block
- Caudal epidural steroid injection group (Active Comparator): Fluoroscopy-guided caudal epidural steroid injection is applied to patients in this group.
  Interventions: Procedure: Fluoroscopy-guided caudal epidural steroid injection

INTERVENTIONS:
Procedure: Fluoroscopy-guided ganglion impar block — Fluoroscopy guidance is used for correct visualization of injection site, and so obtained more successful results. Patients are placed in the prone position. Injection site is cleaned thrice with povidone iodine %10 solution and covered with sterile drapes. Being most commonly used technic, transsacrococcygeal technique, a 22-gauge, 1.5-inch spinal needle is advanced through the sacrococcygeal disk and positioned carefully anterior to the sacrococcygeal junction. Injection of contrast results in a classical comma sign. A mixture of steroid and local anesthetic is given.
  Arms: Ganglion impar block group
Procedure: Fluoroscopy-guided caudal epidural steroid injection — Fluoroscopy guidance is used for correct visualization of injection site, and so obtained more successful results. Patients are placed in the prone position. Injection site is cleaned thrice with povidone iodine %10 solution and covered with sterile drapes. An 18-gauge epidural needle (Tuohy) is advanced at an angle of 45° to the skin until a 'give-way' sensation is felt and position of the needle is confirmed by lateral and anteroposterior fluoroscopic images. Then 5 ml of iohexol solution is injected through it to confirm the position. A properly placed needle would produce a classical 'inverted fern tree' appearance in anteroposterior view after dye injection or a 'filling defect'. The needle is introduced up to S3 level for proper spread of the drug. A mixture of steroid and local anesthetics is given.
  Arms: Caudal epidural steroid injection group

SUMMARY:
Coccygodynia is a disabling pain in the coccyx exacerbated by sitting or rising from sitting. The pain is often pulling or lancinating in quality, may radiate to the sacrum or buttock, and may coexist with lower back pain. Contributing of many physiologic and psychological factors to its etiology, it may be traumatic or idiopathic in origin. Many risk factors are known such as trauma, female gender and obesity. Despite the identification of chronic coccygeal pain hundreds of years ago, its treatment can be difficult and sometimes controversial because of the multifactorial nature of coccygeal pain. Most cases of coccygodynia resolve within weeks to months with or without conservative treatment, but for a few patients, the pain can become chronic and debilitating. First-line treatment options include analgesic drugs, cushion, sit baths, and manuel therapy. Interventional procedures for pain management can be applied to patients who have no response to other conservative modalities. Ganglion impar block and caudal epidural steroid injection are two treatment options for chronic coccygodynia and both of them can be applied by guidance of fluoroscopy and ultrasonography. Radiofrequency ablation is the other option for treatment and eventually, surgical intervention can be done for patients who have refractory pain despite other treatments.

Although efficacy of two interventional procedure for chronic coccygodynia, ganglion impar block and caudal epidural steroid injection, has been well known, no study is exist comparing the efficacy of them. We aimed to compare the efficacy of ganglion impar block and caudal epidural steroid injection in chronic coccygodynia.

DETAILED DESCRIPTION:
The main purpose of this prospective study is the compare the efficacy of fluoroscopy-guided ganglion impar block and caudal epidural steroid injection in patients with chronic coccygodynia. Patients with chronic coccygeal pain are randomly divided into two groups based on the type of the interventional procedure: Group A, fluoroscopy-guided ganglion impar block group and, group B, fluoroscopy-guided caudal epidural steroid injection group. The patients who have chronic coccygeal pain not responding to other conservative treatments will be recruited from physical medicine&rehabilitation and pain medicine outpatient clinics. Detailed information including all aspects of interventional procedures will be given to patients, and inform consent will be obtained. Pain severity will be assessed using Numerical Rating Scale (NRS) as primary outcome. Quality of life and neuropathic pain component will be evaluated with Short Form-12 (SF-12) Questionnaire and Leeds Assessment of Neuropathic Symptoms&Signs Pain Scale (LANSS) as secondary outcomes, respectively. All assessments will be done at pre-interventional period, three weeks and three months after the procedure, with the exception of NRS, it will be also assessed at first hour post-procedure. All assessments will be done by clinician blinding the treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic coccygodynia between the ages of 18 and 65
* Intractable pain over the coccyx despite conservative treatment

Exclusion Criteria:

* History of ganglion impar blockade and/or caudal epidural steroid injection carried out in the last 3 months
* History of lumbar surgery
* Systemic and/or local infections
* Malignancy
* Bleeding diathesis
* Acute fracture
* Known allergy to contrast material and/or local anesthetic substances
* Known history of any psychiatric disorder
* History of pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Change in pain severity of patients from baseline to each checkpoints | from pre-interventional time to post-interventional 1st hour, 3rd week, 3rd month
  Defining the change in Numeric Rating Scale (NRS) score

SECONDARY OUTCOMES:
Change in number of patients with neuropathic pain from baseline to each checkpoints | from pre-interventional time to post-interventional 3rd week, 3rd month
  Defining the change in number of patients with neuropathic pain using Leeds Assessment of Neuropathic Symptoms and Signs Scale (LANSS)
Change the patient reported quality of life assessment from baseline to each checkpoints | from pre-interventional time to post-interventional 3rd week, 3rd month
  Defining the change in quality of life scores of patients using Short Form 12 Health Survey (SF-12)

CONTACTS AND LOCATIONS:
Overall Officials: Savas Sencan, MD, Principal Investigator — Marmara University
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)